CLINICAL TRIAL: NCT05427539
Title: Feasibility Evaluation of Daily Disposable Toric Soft Contact Lenses Manufactured With an Alternative Hydration Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6482
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Results first posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Ocular Physiology

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized into the (test/control) sequence and wear two different study lens designs (test and control designs) one at a time bilaterally over 2 wear periods.
  Interventions: Device: TEST LENS; Device: CONTROL LENS
- CONTROL/TEST (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized into the (control/test) sequence and wear two different study lens designs (test and control designs) one at a time bilaterally over 2 wear periods.
  Interventions: Device: TEST LENS; Device: CONTROL LENS

INTERVENTIONS:
Device: TEST LENS — AO1DfA manufactured with PG hydration
Device: CONTROL LENS — AO1DfA manufactured with IPA hydration

SUMMARY:
This is a bilateral wear, dispensing, randomized, controlled, double-masked, 2-sequence × 2-period crossover study to evaluate ocular physiology following approximately one week of contact lens wear.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

The subject must:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 39 (inclusive) years of age at the time of screening.
4. By self-report, habitually wear soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 2 days per week during the past month.
5. Possess a wearable pair of spectacles that provide correction for distance vision.
6. In both eyes, have astigmatic refractive error suitable for correction with the toric contact lens powers available in this study:

   1. Sphere powers (DS) -1.50 through -4.00 (inclusive) in 0.25 steps
   2. Cylinder powers (DC) -0.75 and -1.25
   3. Axes (°) 170, 180, 10, 80, 90, 100
7. Have best corrected monocular distance visual acuity of 20/30 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

The submit must not:

1. Be currently pregnant or lactating.
2. Be diabetic.
3. Be currently using any ocular medications or have an ocular infection of any type.
4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
6. Be currently wearing monovision or multifocal contact lenses.
7. Be currently wearing lenses in an extended wear modality.
8. Have a history of strabismus or amblyopia.
9. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
10. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.
11. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
12. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
13. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (6):
- United States (6):
  - VRC, Jacksonville, Florida
  - Maitland Vision Center - North Orlando Ave, Maitland, Florida
  - Sacco Eye Group, Vestal, New York
  - Optometry Group, LLC, Memphis, Tennessee
  - Tyler Eye Associates, Tyler, Texas
  - Botetourt Eyecare, LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 66 subjects were enrolled in this study. Of those enrolled, 65 subjects were dispensed at least one study lens, while 1 subject failed to meet all eligibility criteria. Of those dispensed, 62 subjects completed the study while 3 subjects were discontinued.
Groups:
- Senofilcon A Manufactured With PG Hydration\Senofilcon A Manufactured With IPA Hydration: Subjects randomized to receive the senofilcon A contact lenses manufactured with PG hydration during the first period and senofilcon A manufactured with IPA hydration during the second period.
- Senofilcon A Manufactured With IPA Hydration\Senofilcon A Manufactured With PG Hydration: Subjects randomized to receive the senofilcon A contact lenses manufactured with IPA hydration during the first period and senofilcon A manufactured with PG hydration during the second period.
Period: Period 1
Arm/Group | Senofilcon A Manufactured With PG Hydration\Senofilcon A Manufactured With IPA Hydration | Senofilcon A Manufactured With IPA Hydration\Senofilcon A Manufactured With PG Hydration
Started | 31 | 34
Completed | 29 | 33
Not Completed | 2 | 1
Not completed — Unsatisfactory Lens Fitting due to Test Article | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2
Arm/Group | Senofilcon A Manufactured With PG Hydration\Senofilcon A Manufactured With IPA Hydration | Senofilcon A Manufactured With IPA Hydration\Senofilcon A Manufactured With PG Hydration
Started | 29 | 33
Completed | 29 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- Total: Total Subjects
Arm/Group | Total
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (5.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 8
  White | 57
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes With Grade 3 or Higher Slit Lamp Findings
Description: Slit Lamp Findings (SLF) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). This was performed on each subject eye at every study visit (baseline, unscheduled visits and 1-week follow-up). The data was then dichotomized into two groups. Those with grade 3 or higher and those with grade 2 or lower. The proportion of eyes with SLF with grade 3 or higher was reported.
Time Frame: Up to 1-Week Follow-up
Population: All subjects that were dispensed at least one study lens.
Measure: Number; unit: proportion of eyes
Units Other Than Participants: eyes
Groups:
- Senofilcon A Manufactured With PG Hydration: Subjects that wore the senofilcon A contact lenses manufactured with PG hydration during either the first or second period of the study.
- Senofilcon A Manufactured With IPA Hydration: Subjects that wore the senofilcon A contact lenses manufactured with IPA hydration during either the first or second period of the study.
Arm/Group | Senofilcon A Manufactured With PG Hydration | Senofilcon A Manufactured With IPA Hydration
Number analyzed (Participants) | 64 | 63
Number analyzed (eyes) | 128 | 126
proportion of eyes | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 3-weeks per subject.
Arm/Group | Senofilcon A Manufactured With PG Hydration | Senofilcon A Manufactured With IPA Hydration
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/63
Other Adverse Events (participants affected / at risk) | 0/64 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT05427539/Prot_SAP_000.pdf